CLINICAL TRIAL: NCT01961154
Title: Stepping Down of Asthma Medication in Controlled Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kuopio University Hospital (Other)
Responsible Party: Principal Investigator, Heikki Koskela, Respiratory Physician, Kuopio University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KUH5801124
Record Dates: First submitted 2013-10-09; First posted 2013-10-11 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2016-08

CONDITIONS: Asthma
Keywords: Asthma; medication reduction; asthma exacerbation
MeSH Terms: conditions — Asthma | interventions — Fluticasone-Salmeterol Drug Combination; Budesonide, Formoterol Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Medication reduction (Other): All participants undergo similar type of asthma medical reduction. Thus, there is only one arm.
  Interventions: Drug: Asthma medication reduction

INTERVENTIONS:
Drug: Asthma medication reduction — The asthma medications will be reduced in three steps up to total cessation of asthma drugs or up to asthma exacerbation. First step: Long-acting beta-agonist will be discontinued. The use of inhaled corticosteroids is continued, using the same dosage, preparation, and inhaler as before, for six weeks. Second step: medium to high daily inhaled corticosteroids dose is reduced to low daily dose, for six weeks. Third step: low inhaled corticosteroids dose will be stopped, for six weeks. Before each reduction, saline challenge will be performed.
  Other Names: Seretide, Symbicort

SUMMARY:
Background:

The most common asthma drugs, namely inhaled glucocorticoids (ICS) and long-acting beta-2 sympathomimetic drugs (LABA) carry a risk of adverse effects, some of which being potentially severe. Therefore, current guidelines for asthma management recommend that, after a period of symptom control, a reduction of the dose and cessation of the ICSs and LABAs should be attempted. However, reduction in asthma medications sometimes leads to an exacerbation of asthma. Therefore both physicians and asthmatics are often reluctant to reduce or stop asthma medications and asthma over-medication often occurs. A test that could identify those asthmatics who probably would tolerate asthma medication reduction would be useful.

Objectives:

1. To investigate whether airway responsiveness to hypertonic saline can predict the outcome of asthma treatment reduction in subjects with controlled asthma.
2. To get an estimate about how large a proportion of Finnish asthmatic patients use their medications with unnecessarily high doses or would even manage well without any asthma medications.

Study hypothesis:

1. Airway responsiveness to hypertonic saline can predict the outcome of asthma treatment reduction
2. Most of the Finnish asthmatic patients use their medications with unnecessarily high doses

Methods:

This is a prospective study in which the physician responsible for the subject management and medications is blinded from the saline challenge results and the nurse performing the saline challenges is blinded from medications 70 asthmatic patients with both inhaled ICS and LABA will be recruited. Asthma must be well controlled (Juniper's Asthma Control Questionnaire score equal or less than 0.75 ).

The asthma medications will be reduced in three steps, in six weeks' intervals, up to total cessation of asthma drugs or up to asthma exacerbation. The criteria for asthma exacerbation are strictly defined. First step: LABA will be discontinued. The ICS is continued. Second step: medium to high daily ICS dose is reduced to low daily dose. Third step: The low ICS dose will be stopped. Before each reduction, saline challenge will be performed. Asthma diary is kept throughout the study and the subjects will be provided a direct telephone number to a respiratory physician during all hours of day.

DETAILED DESCRIPTION:
Stepping down of asthma medication in controlled asthma

Principal investigator:

Heikki Koskela, MD. Kuopio University Hospital, Unit for Medicine and Clinical Research, Division of Pulmonary Medicine

The study will be started during the year 2012 and will continue for 36 months.

Background

In Finland, asthma is the second most important disorder justifying special reimbursement of asthma medication, thus causing large expenses to the society.

Inhaled corticosteroids (ICS) are the mainstay of modern asthma therapy. When a medium-dose ICS fail to achieve asthma control, they can be combined with long-acting B2-agonist bronchodilators (LABA). Unfortunately, potential side effects of ICSs and LABAs are common with increased frequency with increased dozing. The most common side effects of ICS are benign, like sore and dry throat but also include serious adverse effects like growth retardation in children and adrenal insufficiency. LABAs, in turn can increase the risks of severe asthma exacerbations and even asthma-related deaths. Therefore, current guidelines for asthma management recommend that, after a period of symptom control, a reduction of the dose and cessation of the ICSs and LABAs should be attempted. There are two recommend strategies: The international Global initiative for asthma (GINA) guideline recommends reduction of the ICS dose first, with subsequent LABA cessation. On the contrary, the American Food and Drug Administration (FDA) recommends cessation of LABAs first. In the present study we follow the FDA recommendations.

At present there is limited experimental data on the optimal timing, sequence, and magnitude of treatment reductions in asthma. Usually, the decision for treatment reduction is based on the absence of symptoms for a certain period of time. However, even asthmatic subjects with minimal symptoms may suffer from asthma exacerbation after treatment reduction. Consequently, both physicians and asthmatics are often reluctant to reduce or stop asthma medications. Very probably this is a major reason for the fact that a great proportion of asthmatic subjects use unnecessarily high doses of asthma medications and multiple preparations. For example, in Finland combination preparations containing both LABA and ICS are more commonly prescribed than preparations containing only ICS (Finnish Social Insurance Institution statistics 2010). Very probably many asthmatics would do well even without any asthma medications: In an Italian study with stable asthmatics, all asthma medication could be stopped in 73 % of the subjects.

There has been a great interest to find a biomarker that could identify asthmatic subjects that would tolerate treatment reduction without exacerbation and those in whom the reduction should not be tried. The following biomarkers have been evaluated to predict asthma exacerbation after ICS dose reduction/cessation: Airway challenges with histamine, mannitol, hypertonic saline, and adenosine as well as measurements of exhaled nitric oxide and sputum eosinophils. In adult subjects, the hypertonic airway challenges (mannitol, hypertonic saline) and the adenosine challenge have usually performed best in this respect. However, none of these biomarkers have been able to predict the outcome of the ICS treatment reduction accurately enough to become part of the clinical routine. To our knowledge, there are no studies that have tried to predict asthma exacerbation after LABA cessation.

Hypertonic airway challenges have long been used to assess airways' tendency to constrict in response to external stimuli (=airway responsiveness). Asthmatic subjects are well known to be hyperresponsive to the bronchoconstrictive effect of hypertonic aerosols. During the recent years we have shown that asthmatic subjects are hypersensitive also to the cough-provoking effect of hypertonic aerosols. Furthermore, treatment with ICS decreases the sensitivity to the cough-provoking effect of hypertonic aerosols. Among asthmatics, cough responsiveness to hypertonic saline correlates closely with a well validated asthma control questionnaire. The bronchoconstrictive response and the cough response to hypertonicity are two separate phenomena and therefore provide additional information about the state of the subject's airways. The two responses can be measured during a single challenge.

The cough response to hypertonic aerosols has never been evaluated whether it can predict the outcome of asthma treatment reduction in subjects with stable asthma. It is possible that analysis of both the bronchoconstrictive and the cough response might predict the asthma exacerbation better than analysis of only one of the responses.

The study objectives

Subjects: 70 well-controlled asthmatic patients with both LABA and ICS.

The main objectives of the study:

1. To investigate whether hypertonic saline bronchoconstrictive responsiveness can predict the outcome of asthma treatment reduction in subjects with stable asthma.
2. To investigate whether hypertonic saline cough responsiveness can predict the outcome of asthma treatment reduction in subjects with stable asthma.
3. To investigate whether the two responses together have a stronger predictive power than the responses separately.

The secondary objective is to get an estimate about how large a proportion of Finnish stable asthmatic patients use their medications with unnecessarily high doses or would even manage well without any asthma medications.

Methods

Study design

This is a prospective study in which the physician responsible for the subject management and medications is blinded from the saline challenge results and the nurse performing the saline challenges is blinded from medications. The study includes two periods: A two-week run-in period during which the subjects continue their regular asthma medications and their asthma control is ensured. After that, the stepping down of the asthma medication is started and continued until both ICS and LABA treatments have been stopped or until asthma exacerbation has occurred. The effect of every reduction is observed for six weeks before proceeding to the following step. If the medication is insufficient, an asthma exacerbation is very likely to take place within this time period. In previous studies, the exacerbations have taken place mean 16 - 17 days after steroid reduction.

First step: LABA will be discontinued. The use of ICS is continued, using the same dosage, preparation, and inhaler as before.

Second step: In subjects with a daily ICS dose of more than 500 ug of beclomethasone or equivalent (="medium to high dose"), the ICS dose is reduced to 500 ug of beclomethasone or equivalent ( = "low daily dose") according to GINA, see table 1. The reduced ICS dose will be administered with the same preparation and inhaler as before.

Third step: In subjects with a daily ICS dose of less or equal to 500 ug of beclomethasone or equivalent ( = "low daily dose") the ICS will be stopped.

Non-permitted medications

The use of any asthma drug apart from ICS and LABAs can be continued throughout the study. However, on the study days the subject should not use any asthma drugs before the visit to the outpatient clinic. All medications to other illnesses will be continued throughout the study.

Detailed description of the study

Day 1. The subject will be interviewed (nurse) and the baseline questionnaire and asthma control questionnaire 19 will be filled in. The suitability of the subject for the study is evaluated according to the above-mentioned criteria. Written, informed consent is obtained. If skin allergy tests have not been performed before, it will be performed now. The use of asthma diary is instructed. It will be used throughout the study. A two-week diary monitoring with PEF values will be performed.

Asthma diary:

Every morning and evening: The number of rescue bronchodilating drug doses taken. Three peak flow (PEF) recordings before taking any asthma medication.

Plus every morning: Awakenings at night due to asthma symptoms

Day 2. The diary will be reviewed (physician). The subject will be included in the study if his/her asthma is well controlled, defined as asthma control questionnaire (ACQ) score equal or less than 0.75. The final ACQ score can be determined after the saline challenge since it includes spirometry and forced expiratory volume in one second (FEV1) information is utilised when calculating the ACQ score. If the subject is included, a written asthma medication reduction plan is made, one copy is given to the subject and another is stored in the subject file. The threshold value for significant PEF reduction is calculated (see below). The subject is told about the signs and symptoms of asthma exacerbation and an action plan is made. The saline challenge will be performed (nurse) as described below. The first step-down in the medication is performed (LABA cessation).

Definition of asthma exacerbation, at least one of the following:

* awakening at two consecutive nights due to asthma symptoms
* PEF less than 3 standard deviations from the mean PEF value obtained during the run-in period on three consecutive days 20
* bronchodilator use more than once a day on three consecutive days.
* whenever the subjects feels that his/her asthma symptoms have clearly increased

Individually adjusted definition of asthma exacerbation is written in the asthma diary

Action plan in case of exacerbation: The telephone numbers of the study physicians are given to the subject and she/he can contact them during the office hours. The telephone number of the respiratory physician in charge is given in case of an exacerbation occurring outside the office hours. The exacerbation will be treated according to the standard clinical practice, depending on the physician's judgement. An asthma exacerbation indicates end of the study. The contacted physician informs the research nurse about the exacerbation. The nurse marks down the date of exacerbation. The research nurse asks the patient to visit the outpatient clinic after two weeks. The subject will visit the study physician and the permanent asthma medication will be instructed.

Action plan is written in the asthma diary

Days 3, 4 and 5. The ACQ will be filled in and the diary will be reviewed (physician). If no exacerbations have occurred since the last step-down, the next step-down is made. The hypertonic saline challenge will be performed (nurse). However, if the previous step-down was steroid cessation, the study ends.

Hypertonic saline challenge

This test will be performed as we have previously described with some modifications: Spirometry is performed three times. After that the subject inhales isotonic phosphate-buffered saline for two minutes via a high-output ultrasonic nebuliser, using tidal breathing. The coughs occurring during the inhalation and two minutes after it will be counted up. The number of these "spontaneous" coughs will be subtracted from the coughs provoked by each hypertonic solution. After two minutes from the end of inhalation, the spirometry will be performed twice. The better of the two recorded FEV1 values will be used as the reference value when calculating the saline-induced bronchoconstriction. Subsequently, they inhale hypertonic phosphate-buffered saline solutions with osmolalities of 600, 900, 1200, 1500, 1800 and 2100 milliosmoles (mOsm) /kg. The challenge will be stopped if either if a 15 % fall in FEV1 is recorded or if the final solution has been inhaled or if the patient feels severe discomfort. The cough response to saline will be calculated as the provocative osmolality to induce 15 cumulative coughs. The bronchoconstrictive response will be calculated as the provocative osmolality to induce 15 % fall in FEV1. If the patient feels dyspnoea or if the FEV1 falls equal or more than 15 % from baseline, Ventoline Evohaler two doses a 0.1 mg /Volumatic will be administered. After 15 minutes from that, spirometry will be performed twice.

Ethics

According to international studies, asthma patients often overmedicate themselves, thus being exposed to unnecessary side effects and expenses. Also, due to the vast amount of asthma patients, unnecessary asthma medication causes large expenses to the society. Therefore, the present study is indicated. It is evident that a proportion of the subjects will experience asthma exacerbation during the study. However, they have full-time contact to a respiratory physician. In the study setting, the asthma medication reduction takes place in a much more controlled fashion than in everyday clinical practice.

A permission of the Institutional Ethics Committee has been received (Number 118//2011, dated 29.11.2011).

The time table and financing

The study will be started during the year 2012 and will continue for 36 months. The investigators seek funding from the Finnish government research funding (VTR) and from private foundations.

Investigators and affiliations

Principal investigator: Heikki Koskela, MD, respiratory physician, Kuopio University Hospital, Unit of Medicine and Clinical Research, Department of Respiratory Medicine

Minna Purokivi, MD, respiratory physician, Kuopio University Hospital, Unit of Medicine and Clinical Research, Department of Respiratory Medicine

Jouko Kokkarinen, MD, respiratory physician, Kuopio University Hospital, Unit of Medicine and Clinical Research, Department of Respiratory Medicine

Merja Esselström, registered nurse, MD, Kuopio University Hospital, Unit of Medicine and Clinical Research, Department of Respiratory Medicine

Kirsi Kontra, Pharm. Lic. Kuopio University Hospital, Department of Pharmacy

Analysis of the results, publication plan

The analysis will consist of three parts, one publication will be written about each.

1. The ability of the saline challenge to predict an exacerbation after cessation of LABA will be assessed by comparing the responses to saline between those who tolerated the first reduction (=LABA cessation) and those who did not tolerate it, utilising unpaired T-tests. Suitable cut-off values for saline responses will be sought and after that, the sensitivity and specificity of the saline responses to predict an asthma exacerbation after LABA cessation are defined.
2. The subjects who tolerated the LABA reduction will undergo reductions 2 and 3. The ability of the saline test to predict an exacerbation after reduction/cessation of ICS will be assessed by comparing the results to saline between those who tolerated the second and the third reduction (= ICS reduction and ICS cessation) and those who did not tolerate it, utilising unpaired T-tests. Suitable cut-off values for saline responses will be sought and after that, the sensitivity and specificity of the saline responses to predict an asthma exacerbation after ICS reduction are defined.
3. In addition, the proportion of the subjects who tolerated asthma medication reduction/cessation will be calculated and reported.

ELIGIBILITY:
Inclusion Criteria:70 adult (over 18 years) subjects with the following features

* doctor's diagnosis of asthma and right to special reimbursement from anti-asthma medication expenses according to Finnish Social Insurance Institute criteria (code 203 in the social insurance card)
* asthma diagnosis confirmed at least two years previously
* regular treatment with inhaled corticosteroids and long-acting beta-agonists for at least 6 months
* no changes in regular anti-asthma medication within 6 months
* asthma is well controlled (all conditions must be fulfilled):

  * No courses of oral corticosteroids due to asthma within one year
  * No hospital admissions due to asthma within one year
  * Juniper's Asthma Control Questionnaire score equal or less than 0.75

Exclusion Criteria:

* the presence of another chronic respiratory disease in addition to asthma. Such diseases include moderate to severe polypotic chronic rhinosinusitis, chronic obstructive pulmonary disease, sarcoidosis, and cystic fibrosis
* presence of severe co-morbidity
* history of smoking more than 10 pack-years
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2012-10; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Asthma exacerbation | six weeks
  Possible asthma exacerbation secondary to asthma medication reduction

SECONDARY OUTCOMES:
The proportion of asthma patients able to reduce their medication | 18 weeks
  The number of participants who tolerated at least one step of medication reduction without exacerbation

CONTACTS AND LOCATIONS:
Locations (1):
- Kuopio University Hospital, Kuopio, KYS, Finland